CLINICAL TRIAL: NCT04891133
Title: European DisCoVeRy for Solidarity: An Adaptive Pandemic and Emerging Infection Platform Trial
Brief Title: EU SolidAct: An Adaptive Pandemic and Emerging Infection Platform Trial
Acronym: Bari-SolidAct
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The trial was stopped prematurely due to external evidence that arose during the study period showing that the IMP, baricitinib, was not effective in the primary study population.
Sponsor: Oslo University Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Epidemiological and Clinical Research Information Network (Other)
Responsible Party: Principal Investigator, Marius Trøseid, Associated professor, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EU SolidAct; 2022-500385-99-00 (Other: European Medicines Agency (CTIS))
Record Dates: First submitted 2021-05-07; First posted 2021-05-18 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Emerging Infectious Disease
MeSH Terms: conditions — COVID-19; Communicable Diseases, Emerging | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Corresponding placebo tablets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active arm (Experimental): 4mg Baricitinib up to 14 days + SoC
  Interventions: Drug: Baricitinib
- Comparator (Placebo Comparator): Matching placebo up to 14 days + SoC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — 4 mg baricitinib (2 tablets of 2 mg) once daily
  Other Names: Olumiant
  Arms: Active arm
Drug: Placebo — 4 mg placebo (2 tablets of 2 mg) once daily
  Arms: Comparator

SUMMARY:
EU SolidAct is a randomized, multifactorial, adaptive platform trial for COVID-19 and emerging infectious diseases and pandemics. The purpose of this study is to evaluate the effect of a range of interventions to improve outcome of patients admitted to hospital with COVID-19. The platform is designed for running phase 2 and phase 3 trials, and with modular data capture (end point/safety data, biobanking, add-on studies) depending on the capacity of participating sites. The study consists of two parts with different primary end points depending on disease stage: EU SolidAct part A includes hospitalized patients with moderate disease, whereas EU SolidAct part B includes hospitalized patients with severe and critical disease.

DETAILED DESCRIPTION:
There is an urgent need for developing an adaptive pan-European research platform for rapid and coordinated investigation of new candidate drugs during ongoing pandemics. EU-SolidAct is an Adaptive Platform Trial master protocol developed for evaluating drug interventions in hospitalized patients with COVID-19. While this master protocol is developed for therapeutic interventions in hospitalized patients, it could also form the basis for trial protocols on other interventions and/or in non-hospitalized populations. The protocol is additionally developed to facilitate a joint European response to the challenge of evaluating interventions during future epidemics. The described disease states and endpoints may need to be adapted to the epidemic in question.

EU-SolidAct is a European, multicentre, randomized, parallel, phase 2 and 3 platform trial on drug interventions, both new and repurposed, single or in combination, in hospitalized adult patients with moderate or severe COVID-19, as defined by the WHO Working Group on the Clinical Characterisation and Management of COVID-191. Participants with moderate disease (WHO score 4-5) will be eligible for EU-SolidAct Part A, whereas participants with severe/critical disease (WHO score 6-9) will be eligible for EU-SolidAct Part B. This might include participants progressing from Part A.

In Part A of phase 3 confirmatory trials, the primary objective is to determine the effect of therapeutic interventions on occurrence of disease progression, from moderate disease to severe/critical disease or death within 14 days. In Part B, the primary objective is to determine the effect of therapeutic interventions on occurrence of death within 60 days.

In phase 2 the default objective for both parts is to explore the effect of the therapeutic intervention on respiratory dysfunction at day 5. Other objectives, e.g. effect on virological outcomes may be considered based on the treatment mode of action.

In phase 3 trials, both superiority and non-inferiority hypotheses may be evaluated. In phase 2 trials, only superiority hypotheses will be evaluated. In addition to single treatments, combination of treatments could also be assessed through factorial design. EU-SolidAct is designed to be adaptive and to enable inclusion of hospitals in Europe and beyond, regardless of epidemic waves and available resources. This requires the master protocol to be modular, ranging from a core set of outcomes to more advanced data capture. Hospitals will access the study on different pre-set levels, ranging from a core set of clinical endpoints and safety measures, to a more advanced level with biobanking and possibilities for add-on studies

ELIGIBILITY:
**EU SOLIDACT PLATFORM INCLUSION CRITERIA**:

Participants are eligible to be included in the study only if all the following general inclusion (GI) criteria apply:

* GI1. ≥ 18 years of age
* GI2. Laboratory-confirmed SARS-CoV-2 infection (new infection or reinfection) as determined by PCR not more than 14 days old.
* GI3. Admitted to hospital
* GI4. Informed consent by the participant or legally authorized representative
* GI5A (SolidAct part A): Moderate disease state defined as hospitalised patients without oxygen therapy or oxygen by mask or nasal prongs needed, or
* GI5B (SolidAct part B): Severe/critical disease state defined as fulfilling at least one of the following criteria:

  1. SpO2<90% on room air, or
  2. SpO2 90-94% with a downwards trend and/or signs of respiratory distress*, or
  3. Need of oxygen by NIV (CPAP, BIPAP), high flow or non-rebreather mask, or
  4. Need of mechanical ventilation/ECMO

     * persistently increased respiratory rate, use of accessory muscles, inability to complete full sentences. Clinical judgement must be applied to determine whether a low oxygen saturation is indicative of disease progression or severity or is habitual for a given patient (i.e., with underlying chronic lung disease).

NIV=non-invasive ventilation. CPAP= Continuous Positive Airway Pressure, BPAP= Bi-level Positive Airway Pressure, ECMO = extracorporeal membrane oxygenation.

Additional inclusion criteria are given in the intervention-specific sub-protocols.

Note: these are based on the same criteria as in the WHO living guidelines recommending corticosteroid treatment for severe and critical COVID-195.

In addition, the following specific inclusion criteria apply:

SI-01. Immunocompromised patients defined as the presence of at least one of the following conditions9:

1. Hematological malignancy or pre-malignancy, except acute leukemia or history of lymphoma
2. Organ transplant recipients, except recipients of bone marrow or solid organ transplant last 6 months, or with transplant rejection last 6 months
3. HIV positive with CD4 count < 350 cells and on stable antiretroviral therapy
4. Primary immunodeficiency
5. Rheumatoid arthritis, lupus, vasculitis, inflammatory bowel disease or other autoimmune disorder for which a patient is being treated with systemic immunosuppressive medication
6. Other specified cause, such as history of cancer, cancer treatment or other condition that in the opinion of the investigator could cause impaired host immunity

SI-02. Elevation of 2 or more inflammatory markers above the following cutoffs:

* Ferritin > 700 ug/l
* LDH > 400 U/L
* CRP > 75 mg/L

Note: Carefully check exclusion criteria SE-01, SE-20 and SE-21 (immunosuppressive therapy), SE-22 (medical condition), SE-13 (neutropenia) and SE-14 (lymphopenia) for eligibility criteria.

Immunocompromised patients should receive appropriate SoC, including anti-SARS-CoV2 monoclonal antibodies or emerging antiviral treatment, if available and indicated by current treatment guidelines at time of inclusion.

EXCLUSION CRITERIA:

Participants are excluded from the study if any of the following general exclusion criteria (GE) apply:

* GE1. Anticipated transfer to another non-trial hospital within 72 hours
* Additional exclusion criteria, including prohibited medication, confounding trials and details on contraception and pregnancy are given in the intervention-specific sub-protocols

  * SE-01. Patients receiving Janus kinase (JAK) inhibitors (including baricitinib) for any indication at screening.
  * SE-20. Have received tocilizumab or sarilumab for any indication 4 weeks prior to screening.

Note: Tocilizumab as rescue therapy will be allowed in patients with clinical progression after inclusion, see section 6.8 concomitant medication. If tocilizumab or other immunosuppressive rescue therapy is started, IMP should be discontinued.

• SE-21. Patients with recent changes in immunosuppressive therapy that could interfere with the potential effect of baricitinib.

Note: An assessment of the total level of immunosuppression, hematological parameters (SE-13 and SE-14), drug half-lives, drug-drug interactions, and underlying medical conditions (SE-22) must be performed as part of the risk/benefit evaluation.

* Recipients of bone marrow transplant or solid organ transplant last 6 months, or with transplant rejection last 6 months, should not be included.
* Organ transplant recipients receiving triple immunosuppression can only be included if the anti-metabolite (mycophenolic acid or mTOR inhibitor) has been temporarily discontinued per clinical practice10. IMP should be discontinued once triple immunosuppression is restarted.

  * SE-22. Any medical condition that in the opinion of the investigator poses an inacceptable risk of serious infection or aggravation of the medical condition by participating in the trial.

Note: Patients with acute leukemia or history of lymphoma should not be included. Cancer patients under active treatment, HIV positive individuals with detectable HIV-RNA, or other patient group associated with high risk of serious infection or aggravation of the medical condition should only be included if, in the judgement of the investigator, the potential benefit outweighs the potential risk.

* SE-03. Have received dexamethasone 6 mg daily (or alternative regimens with equivalent of corticosteroids) for more than 4 days prior to screening as part of SoC for severe/critical COVID-19
* SE-04. Had COVID-related symptoms > 21 days or hospitalized > 7 days.
* SE-05. Strong inhibitors of organic anion transporter 3 [OAT3] (e.g., probenecid) that cannot be discontinued at study entry.
* SE-07. Have received any live vaccine within 4 weeks before screening, or intend to receive a live vaccine during the study (until day 90 (+/- 14 days)).

Note: Use of non-live (inactivated) vaccinations, including COVID-19 vaccinations, is allowed for all participants.

* SE-08. Are using or will use extracorporeal blood purification (EBP) device to remove proinflammatory cytokines from the blood such as a cytokine absorption or filtering device, for example, CytoSorb®.
* SE-09. Have diagnosis of current active tuberculosis (TB) or, if known, latent TB treated for less than 4 weeks with appropriate anti-tuberculosis therapy per local guidelines (by history only, no screening tests required).
* SE-10. Suspected serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking investigational product.
* SE-12. Have a history of venous thromboembolism (VTE) (deep vein thrombosis [DVT] and/or pulmonary embolism [PE]) within 12 weeks prior to randomization or have a history of recurrent (>1) VTE (DVT/PE).
* SE-13. Neutropenia (absolute neutrophil count <1000 cells/microliters).
* SE-14. Lymphopenia (absolute lymphocyte count <200 cells/microliters).
* SE-15. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 times ULN.
* SE-16. Subjects with estimated glomerular filtration rate (eGFR) (Modification of Diet in Renal Disease [MDRD]) <30 millilitre/minute/1.73 meters squared are excluded.
* SE-17. Known hypersensitivity to baricitinib or any of its excipients.
* SE-18. Are pregnant or breastfeeding, or intend to become pregnant or breastfeed during the study.

Note: Women of child bearing potential (WOCBP) can only be included based on a negative pregnancy test and WOCBP must comply with requirements regarding highly effective contraception. Refer to section 10.1 for contraception requirements.

• SE-19 Participation in any therapeutic clinical trials investigating immunomodulators for COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Occurrence of death within 60 days (primary end point, EU SolidAct part B) | 60 days
  The primary outcome for phase 3 trials in EU SolidAct part B is occurrence of death within 60 days
Occurrence of disease progression within 14 days (primary end point, EU SolidAct part A) | 14 days
  The primary outcome for phase 3 trials in EU SolidAct part A is occurrence of disease progression, defined as a progression of disease state from moderate (WHO score 4-5) to severe/critical (WHO score 6-9) or death (WHO score 10)
SpO2/FiO2-ratio at day 5 (primary end point, phase 2 trials) | 5 days
  In phase 2 exploratory trials, the default primary objective for both part A and B is to explore the effect of the intervention on respiratory dysfunction assessed by SpO2/FiO2-ratio at day 5

SECONDARY OUTCOMES:
Occurrence of disease progression within 28 days (shared secondary end point for part A and B) | 28 days
  Occurrence of disease progression, defined as a progression of disease state from moderate (WHO score 4-5) to severe/critical/death (WHO score 6-10) or from severe/critical (WHO score 6-9) to death
Time to sustained recovery (shared secondary end point for part A and B) | 90 days
  Time from randomization to sustained recovery, defined as being discharged from the index hospitalization, followed by being alive and at home for 14 consecutive days within 90 days
Time to first hospital discharge (shared secondary end point for part A and B) | 90 days
  Time from randomization to first hospital discharge within 90 days
Disease state at Day 15 and Day 29 (shared secondary end point for part A and B) | 28 days
  Disease state on a 5-point scale defined as:
  1. Mild (WHO score 1-3) or better,
  2. Moderate (WHO score 4-5),
  3. Severe (WHO score 6),
  4. Critical (WHO score 7-9) or
  5. Death at Day 15 and 29
Time from randomization to recovery (shared secondary end point for part A and B) | 90 days
  Time from randomization to recovery defined as no need for oxygen
SpO2/FiO2-ratio at Day 3, 5 and 8 (shared secondary end point for part A and B) | 8 days
  Respiratory dysfunction assessed by SpO2/FiO2-ratio at Day 3, 5 and 8
Viral clearance during hospitalization (shared secondary end point for part A and B) | Days 1, 3, 5, 8 and 15
  Viral clearance as assessed by SARS-CoV-2 PCR in naso/oropharyngeal specimens collected at Days 1, 3, 5, 8 and 15 (± 1 day, except baseline) if still hospitalized
Occurrence of serious adverse events within 90 days (shared secondary end point for part A and B) | 90 days
  Occurrence of serious adverse events leading to study treatment discontinuation or death
Patient related outcomes at day 90 (shared secondary end point for part A and B) | 90 days
  The Oslo COVID-19 QLQ-PW80 subscale scores at Day 90

OTHER OUTCOMES:
Changes in C-reactive protein from baseline | Days 1, 3, 5, 8, 15 and 22
  Analyzed in blood samples collected at Days 1, 3, 5, 8, 15 and 22 (± 1 day) if still hospitalized
Changes in Ferritin from baseline | Days 1, 3, 5, 8, 15 and 22
  Analyzed in blood samples collected at Days 1, 3, 5, 8, 15 and 22 (± 1 day) if still hospitalized
Changes in Lactate dehydrogenase from baseline | Days 1, 3, 5, 8, 15 and 22
  Analyzed in blood samples collected at Days 1, 3, 5, 8, 15 and 22 (± 1 day) if still hospitalized
Changes in D-dimer from baseline | Days 1, 3, 5, 8, 15 and 22
  Analyzed in blood samples collected at Days 1, 3, 5, 8, 15 and 22 (± 1 day) if still hospitalized
Changes in procalcitonin from baseline | Days 1, 3, 5, 8, 15 and 22
  Analyzed in blood samples collected at Days 1, 3, 5, 8, 15 and 22 (± 1 day) if still hospitalized
Changes in neutrophils from baseline | Days 1, 3, 5, 8, 15 and 22
  Analyzed in blood samples collected at Days 1, 3, 5, 8, 15 and 22 (± 1 day) if still hospitalized
Changes in lymphocytes from baseline | Days 1, 3, 5, 8, 15 and 22
  Analyzed in blood samples collected at Days 1, 3, 5, 8, 15 and 22 (± 1 day) if still hospitalized
Changes in White Blood Cell Count from baseline | Days 1, 3, 5, 8, 15 and 22
  Analyzed in blood samples collected at Days 1, 3, 5, 8, 15 and 22 (± 1 day) if still hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Domique Costagliola, PhD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France; Jose R Arribas, MD PhD, Principal Investigator — Hospital Universario La Paz, Madrid
Locations (92):
- Austria (3):
  - Medical University of Innsbruck (University Hospital for Neurosurgery), Innsbruck
  - Medical Unversity of Innsbruck (Joint Institute for Emergency Medicine and Critical Care), Innsbruck
  - Medical Unversity of Innsbruck (University Hospital for Anaesthesia and Intensive Care), Innsbruck
- Belgium (3):
  - Erasme Hospital, Brussels
  - UZ Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
- St Anne University Hospital, Brno, Czechia
- France (16):
  - CHU Amiens Picardie (ICU), Amiens
  - CHU Amiens Picardie (ID), Amiens
  - CHU de Bordeaux / Hopital Pellegrin (ICU), Bordeaux
  - CHU de Bordeaux / Hopital Pellegrin (ID), Bordeaux
  - Louis Mourier (ID), Colombes
  - Lous Mourier (ICU), Colombes
  - CHU François Mitterrand, Dijon
  - CHU Lille - Hopital Roger Salengro -Pôle Rèanimaition, Lille
  - Hopital de la Croix - Rousse - HCL (ICU), Lyon
  - Hopital de la Croix - Rousse - HCL (ID), Lyon
  - GHRMSA Hopital Emile Muller (ICU), Mulhouse
  - GHRMSA Hopital Emile Muller (IM), Mulhouse
  - Hôpital Saint-Antoine (ICU), Paris
  - Hôpital Saint-Antoine (ID), Paris
  - Hôpital Bichat - Claude Bernard (ICU), Paris
  - Hôpital Bichat - Claude Bernard (ID), Paris
- Germany (2):
  - Gesundheit Nord gGmbH (GeNo), Bremen
  - Technische Universität München (TUM) - Klinikum rechts der Isar, München
- Greece (2):
  - Evangelismos Hospital, Athens
  - Attikon University Hospital, Athens
- Hungary (3):
  - University of Debrecen (Clinic for Infectology), Debrecen
  - University of Pécs, Pécs
  - University of Szeged (Pandemic Clinics), Szeged
- Ireland (8):
  - Cork University Hospital, Cork
  - St Vincent's University Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St James's Hospital, Dublin, Dublin
  - Beaumont Hospital, Dublin, Dublin
  - Tallaght University Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Limerick, Limerick
- Italy (17):
  - Ospedale Santa Maria Annunziata, Malattie Infettive, Bagno a Ripoli
  - ASST - Spedali Civili di Brescia - University of Brescia, Brescia
  - ATS Sardegna - PO SS Trinità, U.O.C. Malattie Infettive, Cagliari
  - Azienda Opsedaliera Universitaria Mater Domini, U.O. Malattie Infettive e Tropicali, Catanzaro
  - ASL Frosinone - Ospedale Fabrizio Spaziani, U.O.C. Medicina Interna, Frosinone
  - Ospedale S.M. Goretti di Latina, U.O.C. Malattie Infettive, Latina
  - Ospedale Mater Salutis di Legnago, U.O.C. di Pneumologia, Legnano
  - Ospedale Mater Salutis di Legnago, U.O.S. di Malattie Infettive, Legnano
  - ASST Santi Paolo e Carlo, S.C. Malattie Infettive, Milan
  - Azienda Ospedaliera Universitaria Vanvitelli, U.O.C. Malattie Infettive, Napoli
  - AOU Policlinico "P. Giaccone", U.O.C. Malattie Infettive, Palermo
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, U.O.C. Malattie Infettive, Pesaro
  - ASL Taranto - Ospedale Oncologico San Giuseppe Moscati, U.O.C. Pneumologia, Taranto
  - AOU Città della Salute e Scienza Presidio Molinette, Torino
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI), S.C. Malattie Infettive, Trieste
  - IRCCS Ospedale Sacro Cuore Don Calabria, U.O.S. Malattie Infettive e Tropicali, Verona
  - Azienda Ospedaliera Universitaria Integrata di Verona, U.O.C. Malattie Infettive e Tropicali, Verona
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Norway (10):
  - Drammen (Vestre Viken) Hospital, Drammen
  - Østfold sykehuset i Kalnes, Grålum
  - Akershus Universitetssykehus, Lørenskog
  - Lovisenberg Diaconal Hospital, Oslo
  - OUS Ullevål, Oslo
  - Bærum Hospital, Sandvika
  - Stavanger University Hospital, Stavanger
  - University Hospital North Norway, Tromsø
  - St. Olavs Hospital, Trondheim
  - Vestfold Hospital, Tønsberg
- Portugal (8):
  - CHMT - Centro Hospitalar do Médio Tejo- Hospital de Abrantes, Abrantes
  - CHUC - Centro Hospitalar e Universitário de Coimbra, Coimbra
  - CHUA-Faro - Centro Hospitalar Universitário do Algarve, Faro
  - CHLC-HCC - Hospital Curry Cabral, Centro Hospitalar Universitário Lisboa Central, Lisbon
  - CHLO - Centro Hospitalar de Lisboa Ocidental - HEM and HSFX, Lisbon
  - CHSJ - São João Hospital Center, Lisbon
  - CHLN - Centro Hospitalar Universitário Lisboa Norte, Lisbon
  - HBA - Hospital Beatriz Ângelo, Loures
- Slovakia (5):
  - University Hospital Bratislava, Kramare, Bratislava
  - University Hospital Martin, Martin
  - Nsp Trebisov, Svet Zdravia a.s., Trebišov
  - Faculty Hospital Trencin, Trenčín
  - University Hospital Trnava, Trnava
- Spain (8):
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Jaen, Jaén
  - Hospital Universitario La Paz, Madrid
  - Hospital Costa del Sol, Marbella
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen de Valme, Seville
- Turkey (Türkiye) (5):
  - Hacettepe Üniversitesi Tıp Fakültesi, İnfeksiyon Hastalıkları ve Klinik Mikrobiyoloji Anabilim Dalı (Site 1), Ankara
  - Hacettepe Üniversitesi Tıp Fakültesi, İnfeksiyon Hastalıkları ve Klinik Mikrobiyoloji Anabilim Dalı (Site 2), Ankara
  - Ankara Üniversitesi Tıp Fakültesi, Enfeksiyon Hastalıkları ve Klinik Mikrobiyoloji Anabilim Dalı, Ankara
  - İstanbul Üniversitesi İstanbul Tıp Fakültesi, Enfeksiyon Hastalıkları ve Klinik Mikrobiyoloji Anabilim Dalı, Istanbul
  - Dokuz Eylül Üniversitesi Tıp Fakültesi Enfeksiyon Hastalıkları ve Klinik Mikrobiyoloji Anabilim Dalı, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Individual patient-level data will be made as public as possible while maintaining the integrity and privacy of the trial participants. Anonymized data will be made publicly available using a data repository, including any programming code used to produce the trial results. De-identified data will be made available upon request and evaluation of the requestee's ability and willingness to maintain the integrity and privacy of the trial participants. Further details of data sharing will be given in a separate data sharing plan.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Troseid M, Arribas JR, Assoumou L, Holten AR, Poissy J, Terzic V, Mazzaferri F, Bano JR, Eustace J, Hites M, Joannidis M, Paiva JA, Reuter J, Puntmann I, Patrick-Brown TDJH, Westerheim E, Nezvalova-Henriksen K, Beniguel L, Dahl TB, Bouscambert M, Halanova M, Peterfi Z, Tsiodras S, Rezek M, Briel M, Unal S, Schlegel M, Ader F, Lacombe K, Amdal CD, Rodrigues S, Tonby K, Gaudet A, Heggelund L, Mootien J, Johannessen A, Moller JH, Pollan BD, Tveita AA, Kildal AB, Richard JC, Dalgard O, Simensen VC, Balde A, de Gastines L, Del Alamo M, Aydin B, Lund-Johansen F, Trabaud MA, Diallo A, Halvorsen B, Rottingen JA, Tacconelli E, Yazdanpanah Y, Olsen IC, Costagliola D; EU SolidAct study group. Efficacy and safety of baricitinib in hospitalized adults with severe or critical COVID-19 (Bari-SolidAct): a randomised, double-blind, placebo-controlled phase 3 trial. Crit Care. 2023 Jan 10;27(1):9. doi: 10.1186/s13054-022-04205-8. PMID 36627655
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343